CLINICAL TRIAL: NCT02604667
Title: Mechanisms of Ischemic Stroke in Cancer Patients
Acronym: MOST-CA
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: University of California, Davis (Other); Memorial Sloan Kettering Cancer Center (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1411015653; K23NS091395 (NIH)
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Stroke; Cancer
Keywords: Biomarkers; Mechanisms; Transcranial Doppler
MeSH Terms: conditions — Stroke; Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Cancer and Stroke: Patients with active solid tumor cancer and acute ischemic stroke. Will undergo blood tests and transcranial Doppler microemboli detection study.
  Interventions: Other: Blood tests; Other: Transcranial Doppler Microemboli Detection Study
- Group 2: Stroke and No Cancer: Patients with acute ischemic stroke and no cancer. Will undergo blood tests and transcranial Doppler microemboli detection study.
  Interventions: Other: Blood tests; Other: Transcranial Doppler Microemboli Detection Study
- Group 3: Cancer and No Stroke: Patients with active solid tumor cancer and no stroke. Will undergo blood tests and transcranial Doppler microemboli detection study.
  Interventions: Other: Blood tests; Other: Transcranial Doppler Microemboli Detection Study

INTERVENTIONS:
Other: Blood tests — Study participants will undergo a single, peripheral blood draw. Blood specimens will be used to perform hematological biomarker testing and leukocyte RNA gene expression analysis.
  Hematological biomarker testing will be performed to better elucidate the mechanisms of ischemic stroke in cancer patients and will include markers of coagulation, platelet function, and endothelial integrity. This analysis will occur at MSKCC.
  Leukocyte RNA gene expression analysis will be performed to evaluate whether patients with cancer and stroke more often have cardioembolic mechanisms than patients with stroke and no cancer. This analysis will occur at the University of California, Davis where investigators have previously shown that differential RNA expression patterns can predict stroke subtypes.
Other: Transcranial Doppler Microemboli Detection Study — Study participants will undergo a single Transcranial Doppler Microemboli Detection Study at NYPH/WCMC or MSKCC within two weeks of enrollment. Both middle cerebral arteries will be insonated for 30 minutes by a trained technician or stroke neurologist certified in neurosonology using a fixed headset to assess for the rate and laterality of microemboli.

SUMMARY:
The purpose of this study is to better understand the causes of stroke in people with cancer. Active cancer increases the risk of stroke. The investigators do not know exactly why this occurs but one possible reason is that people with cancer may have thicker blood than people without cancer. Thick blood can sometimes cause blood clots to form in the heart, which can then travel to the brain and cause stroke. This study is being done to help figure out why this and other causes of stroke occur in people with cancer. The investigators expect that information from this study will help doctors to more effectively prevent and treat stroke in individuals with cancer.

DETAILED DESCRIPTION:
This will be a prospective cross-sectional study to examine the unique mechanisms of ischemic stroke in cancer patients. Enrollment will occur at the NewYork-Presbyterian Hospital (NYPH)/Weill Cornell Medical Center (WCMC) and the Memorial Sloan Kettering Cancer Center (MSKCC). Measurements will occur at the NYPH/WCMC and MSKCC Neurovascular Ultrasound Laboratories, the MSKCC Central Laboratory, and the Sharp Laboratory at the University of California, Davis. Three groups of adult patients will be enrolled. Group 1 will consist of consecutive patients with active solid tumor cancer and acute ischemic stroke. Group 2 will be patients with acute ischemic stroke and no cancer. Patients in Groups 1 and 2 will be enrolled at 96 hours +/- 24 hours of stroke onset. Group 3 will include patients with active solid tumor cancer and no stroke. This group will allow us to confirm that differences between stroke patients with and without cancer are not simply incidental findings that can be expected in all cancer patients regardless of thrombotic status. Demographics, comorbidities, and stroke severity (for Groups 1 and 2 only) will be recorded on admission using a structured form. Study patients will undergo three facets of testing: 1) Transcranial Doppler (TCD) microemboli detection; 2) hematological biomarker testing; 3) peripheral blood leukocyte RNA gene expression analysis.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age or older
* Active solid tumor cancer (for Groups 1 and 3 only)
* MRI confirmed acute ischemic stroke (for Groups 1 and 2 only)
* Available for blood draw at 96 hours (+/- 24 hours) from last known well time (for Groups 1 and 2 only) or within 2 weeks of enrollment (for Group 3)
* Available for TCD within 2 weeks of enrollment

Exclusion Criteria

* Primary brain tumor or hematological cancer
* Treatment with intravenous or intraarterial thrombolysis or mechanical embolectomy
* Platelets < 50,000/mm3
* Hemodialysis within 14 days
* Active pregnancy
* Infection within 14 days per Infectious Diseases Society of America (IDSA) criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to enroll three groups of 50 patients each. Group 1 will consist of patients with acute ischemic stroke and active solid tumor cancer, Group 2 will include patients with acute ischemic stroke and no cancer, and Group 3 will include patients with active solid tumor cancer and no stroke.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Hematological biomarker levels | At enrollment
  Hematological testing will consist of a single peripheral blood draw at 96 hours (+/-24 hours). Several factors will be evaluated, including markers of coagulation (thrombin-antithrombin complex, D-dimer), platelet function (P-selectin), and endothelial integrity (sICAM-1, sVCAM-1, thrombomodulin).

SECONDARY OUTCOMES:
Peripheral leukocyte RNA gene expression profiles | At enrollment
  Blood specimens will be collected at the time of enrollment in PAXgene tubes which will be frozen and stored at the Weill Cornell CTSC Core laboratory and sent in batches to the UC Davis laboratory where processing of RNA gene expression will occur.

OTHER OUTCOMES:
Transcranial Doppler microemboli rates | At enrollment
  With TCD studies, both middle cerebral arteries will be insonated for 30 minutes using a fixed headset. An experienced technologist will review the recording to ensure accurate characterization of all signals and a vascular neurologist with expertise in neurosonology will determine the rate and laterality of the microemboli. TCD microemboli in bilateral vascular distributions indicates a central embolic source.

CONTACTS AND LOCATIONS:
Overall Officials: Babak Navi, MD, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Navi BB, Mathias R, Sherman CP, Wolfe J, Kamel H, Tagawa ST, Saxena A, Ocean AJ, Iadecola C, DeAngelis LM, Elkind MSV, Hull H, Jickling GC, Sharp FR, Ander BP, Stamova B. Cancer-Related Ischemic Stroke Has a Distinct Blood mRNA Expression Profile. Stroke. 2019 Nov;50(11):3259-3264. doi: 10.1161/STROKEAHA.119.026143. Epub 2019 Sep 12. PMID 31510897